CLINICAL TRIAL: NCT01290653
Title: Dry Needling Versus Strain Counterstrain Technique: Pilot Study Comparing Effects Over the Upper Trapezius Myofascial Trigger Point
Brief Title: Dry Needling Versus Strain-counterstrain on the Upper Trapezius
Acronym: DNJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, PhD, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU UCH 203
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dry Needling of trigger point (Experimental): Deep dry needling will be applied on the upper trapezius myofascial trigger point
  Interventions: Other: Dry needling
- Strain-counterstraing technique (Experimental): This manual technique will be applied at the upper trapezius.
  Interventions: Other: Strain-counterstrain technique
- Placebo manual technique (Placebo Comparator): A technique simulating strain-counterstrain, but without any therapeutic manoeuvre will be applied at the upper trapezius site.
  Interventions: Other: Placebo manual technique

INTERVENTIONS:
Other: Dry needling — Deep dry needling until achieving twitch response of the muscle
  Arms: Dry Needling of trigger point
Other: Strain-counterstrain technique — A manual technique to release tension of painful muscles.
  Arms: Strain-counterstraing technique
Other: Placebo manual technique — A placebo technique, consisting of manual contact of the therapist with the patient without any further therapeutic approach
  Arms: Placebo manual technique

SUMMARY:
This study investigates the effect of two different techniques (dry needling and Strain-counterstrain manual technique) on the upper trapezius myofascial trigger point (MTP). Subjects with active or latent MTP in this location of the muscle will be identified and will be randomly assigned to one out of three groups: dry needling, strain-counterstrain or placebo manual technique. Pain pressure threshold, provoked pain, pain at rest, neck disability and electromyography (EMG) activity of the upper trapezius will be registered before and after six sessions of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Active myofascial trigger point at the upper trapezius

Exclusion Criteria:

* Diagnosed fibromyalgia
* Cervical radiculopathy
* Facial neuralgia
* Coagulation alteration
* Cancer
* Allergy (included needles)
* History of cervical or shoulder surgery
* History of deep venous thrombosis
* History of myopathy
* History of infiltration at upper trapezius trigger point
* Anticoagulant medication
* Aspirin intake during the last 3 days
* Drug intake (AINES, narcotics, antiepileptics, or any other analgesic medication)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pain Pressure Threshold | 6 sessions
  Amount of pressure (Kg/cm2) applied at the myofascial trigger point site that elicit pain for the patient will be reported. Analogy pressure algometer(Wagner, FPK 20) will be used.

SECONDARY OUTCOMES:
Pain at rest | 6 sessions
  Visual Analogue Scale
Neck Disability | 6 sessions
  Neck Disability Index
Electromyographic activity of the upper trapezius | 6 sessions
  Surface EMG will be recorded (MP 100 de BIOPAC Systems; Goleta, California, USA). Electrodes will be located to register activity of the Upper trapezius, according to Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM) guidelines. Microvolts of activity at rest will be recorded. Data will be normalized through calculation of maximal voluntary contraction, so that final data will be reported as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Segura-Ortí, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain

REFERENCES:
- [Derived] Segura-Orti E, Prades-Vergara S, Manzaneda-Pina L, Valero-Martinez R, Polo-Traverso JA. Trigger point dry needling versus strain-counterstrain technique for upper trapezius myofascial trigger points: a randomised controlled trial. Acupunct Med. 2016 Jun;34(3):171-7. doi: 10.1136/acupmed-2015-010868. Epub 2016 Jan 8. PMID 26746173